CLINICAL TRIAL: NCT03433911
Title: BLOC: Prospective Multi-Center Office Based Bi-Lateral Tubal Occlusion Trial for Female Permanent Contraception
Brief Title: FemBloc® Permanent Contraception - Early Pivotal Trial
Acronym: BLOC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Femasys Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CP-100-007
Record Dates: First submitted 2018-02-01; First posted 2018-02-15 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Contraception
Keywords: Permanent contraception; Birth control

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- FemBloc (Experimental): Investigational device and procedure
  Interventions: Device: FemBloc
- Control (Active Comparator): Laparoscopic bilateral tubal sterilization
  Interventions: Procedure: Laparoscopic bilateral tubal sterilization

INTERVENTIONS:
Device: FemBloc — Treatment with FemBloc for women who desire permanent birth control (female sterilization)
  Arms: FemBloc
Procedure: Laparoscopic bilateral tubal sterilization — Laparoscopic bilateral tubal sterilization for women who desire permanent birth control (female sterilization)
  Arms: Control

SUMMARY:
Prospective, multi-center, international, non-randomized, two-arm study of subjects undergoing either FemBloc or laparoscopic bilateral tubal sterilization (Control). The FemBloc group total study duration will be approximately 65 months. The laparoscopic tubal sterilization (Control) group total study duration will be approximately 62 months.

ELIGIBILITY:
Inclusion Criteria:

* Female, 21 - 45 years of age desiring permanent birth control
* Sexually active with male partner
* For FemBloc Arm:

  * Regular menstrual cycle for last 3 months or on hormonal contraceptives
* For Control Arm:

  * Undergoing planned laparoscopic bilateral tubal sterilization

Exclusion Criteria:

* Uncertainty about the desire to end fertility
* Known or suspected pregnancy
* Prior tubal surgery, including sterilization attempt
* Prior endometrial ablation
* Presence, suspicion, or previous history of gynecologic malignancy
* Abnormal uterine bleeding requiring evaluation or treatment
* Scheduled to undergo concomitant intrauterine procedures at the time of procedure(s)

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of short-term and long-term adverse events in each arm | 1-5 years
  Safety: Incidence of short-term and long-term adverse events in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor, Study Director — Medical Affairs & Clinical Development
Locations (12):
- United States (12):
  - New Horizons Clinical Trials, Chandler, Arizona
  - Stanford University, Stanford, California
  - Altus Research Inc., Lake Worth, Florida
  - Rosemark Womencare Specialists, Idaho Falls, Idaho
  - Women's Health Advantage, Fort Wayne, Indiana
  - Rutgers, The State University of New Jersey, Newark, New Jersey
  - Columbia University Medical Center, New York, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - University Hospitals Cleveland Medical Center, Beachwood, Ohio
  - Amy Brenner MD & Associates, Mason, Ohio
  - Chattanooga Medical Research LLC, Chattanooga, Tennessee
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- See also: FemBloc Study Website — http://www.fembloc.com/